CLINICAL TRIAL: NCT00787059
Title: Phase I/II Study AC6 Gene Transfer for Congestive Heart Failure
Brief Title: AC6 Gene Transfer for CHF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hammond, H. Kirk, M.D. (Individual)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Renova Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 365; P01HL066941 (NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2017-08

CONDITIONS: Congestive Heart Failure
Keywords: Adenylyl Cyclase; AC6; adenovirus; gene therapy; congestive heart failure; intracoronary; nitroprusside
MeSH Terms: conditions — Heart Failure; Adenoviridae Infections | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ad5.hAC6 (Experimental): Will receive intracoronary adenovirus encoding human adenylyl cyclase type 6
  Interventions: Drug: Ad5.hAC6
- sucrose solution (Placebo Comparator): Will receive intracoronary sucrose solution
  Interventions: Drug: Sucrose (3%)

INTERVENTIONS:
Drug: Ad5.hAC6 — Intracoronary delivery of test substance in 3:1 randomization (Ad5.hAC6 : placebo) with dose escalation, starting at 3.2 x 10^9 vp to 10^12 vp in 5 dose groups
  Arms: Ad5.hAC6
Drug: Sucrose (3%)
  Arms: sucrose solution

SUMMARY:
This research study is designed to determine: 1) whether gene transfer using an agent called Ad5.hAC6 (adenovirus-5 encoding human adenylyl cyclase type 6) can be given safely to patients with congestive heart failure (CHF) and 2) whether this agent may be of benefit in heart failure. Gene transfer is a process by which genes are introduced into cells and the cells then produce the specific protein that the gene directs, in this case, a protein known as adenylyl cyclase type 6 (AC6). The gene is carried into the heart cells by a modified virus. The virus that is modified is an adenovirus (Ad5), a virus that sometimes causes a brief cold. In extensive animal experiments, it was found that increased amounts of AC6 protein in heart cells appeared to make the heart pump more vigorously.

DETAILED DESCRIPTION:
This research study is designed to determine: 1) whether gene transfer using an agent called Ad5.hAC6 (adenovirus-5 encoding human adenylyl cyclase type 6) can be given safely to patients with congestive heart failure (CHF) and 2) whether this agent may be of benefit in heart failure. Gene transfer is a process by which genes are introduced into cells and the cells then produce the specific protein that the gene directs, in this case, a protein known as adenylyl cyclase type 6 (AC6). The gene is carried into the heart cells by a modified virus. The virus that is modified is an adenovirus (Ad5), a virus that sometimes causes a brief cold. In extensive animal experiments, it was found that increased amounts of AC6 protein in heart cells appear to make the heart pump more vigorously.

ELIGIBILITY:
Inclusion Criteria

1. Male or non-pregnant female patients aged 18-80 years of age
2. ≥3-month history of heart failure
3. Compensated (stable) CHF not on intravenous inotropes, vasodilators or diuretics, on optimal medical and device therapy as defined by AHA/ACC Guidelines
4. LV ejection fraction (on optimal therapy) no greater than 40%
5. Implanted cardiac defibrillator
6. At least one major coronary artery (or graft) with <50% proximal obstruction
7. Patients unable to walk (spinal injury, orthopedic problems) can be enrolled if all other criteria are met.
8. Women of child-bearing capacity must have a negative pregnancy test within 2 days of test substance administration, and female and male patients must be willing to use birth control during sex for 12w after test substance administration if the female partner is of child-bearing capacity.
9. Subjects willingly provide informed consent consistent with ICH-GCP guidelines

Exclusion Criteria

1. Unstable or Class IV angina
2. Coronary revascularization planned or predicted in next 6 months
3. Ischemic myocardium in 3 or more regions of a single perfusion bed, as assessed by stress echocardiography or jeopardized viable myocardium >15% on perfusion imaging.
4. ≥50% occlusion of an "unprotected" left main coronary artery. If arterial or venous conduits provide blood flow to the distal left coronary circulation (ie, patent bypass grafts) then left main disease is "protected" and such patients are not excluded. The cardiologist performing the cardiac catheterization will make these decisions.
5. 2° AV Block (Mobitz 2) or 3° AV block unless pacemaker is present
6. Hospitalization for CHF requiring intravenous inotropes or vasodilators in the past 4 weeks
7. History of biopsy proven myocarditis
8. Myocardial infarction in previous 6 months
9. Restrictive, hypertrophic or infiltrative cardiomyopathy or chronic pericarditis
10. Previous or planned organ transplant recipient or donor.
11. Thrombocytopenia (<100,000 platelets/µl) or bleeding diathesis
12. COPD requiring supplemental oxygen at home
13. AST > 2 times upper limit of normal or chronic liver disease such as cirrhosis or Hepatitis C Virus (HCV). Patients with HCV are eligible only if both of two conditions are met: a) liver function tests are normal; AND b) liver biopsy is normal or shows only mild fibrosis.
14. Current or predicted hemodialysis within 12 months or estimated glomerular filtration rate (EGFR) <30 ml/min. On online EGFR calculator that uses sex, age, body weight and serum creatinine is available at: www.kidney.org/professionals/kdoqi/gfr_calculator.cfm. Use the higher of two EGFR results, which are based upon MDRD and CKD-EPI formulas.
15. CVA or TIA <6 months prior to enrollment
16. Patients who are immunosuppressed by medicines (corticosteroids, methotrexate, cyclophosphamide, cyclosporine), illnesses (AIDS, HIV), or neutrophil count <1000/mm3
17. Patients receiving other investigational drug therapy within 30 days of enrollment including gene transfer
18. Patients with diseases other than CHF that, in the opinion of the investigator, put the subject at risk or adversely affect the results

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2010-07; Primary Completion 2015-01 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Combined: a) Exercise treadmill time; b) LV function by echocardiography before and during dobutamine infusion; c) Rate of LV pressure development and decline (dP/dt and -dP/dt) before and during dobutamine infusion. | Before, 4w, 12w

SECONDARY OUTCOMES:
Symptoms (KCCQ); hemodynamics; ICD discharge frequency | Before, 4w, 12 w

CONTACTS AND LOCATIONS:
Overall Officials: H. Kirk Hammond, MD, Study Director — UCSD; VA San Diego Healthcare System; Veterans Medical Research Foundation; William Penny, MD, Principal Investigator — UCSD; VA San Diego Healthcare System; Veteran's Medical Research Foundation; Jay H Traverse, MD, Principal Investigator — Minneapolis Heart Institute Foundation; Clyde W Yancy, MD, Principal Investigator — Bluhm Cardiovascular Institute, Northwestern Memorial Hospital; Matthew W Watkins, MD, Principal Investigator — Fletcher Allen Health Care, University of Vermont; Eric D Adler, MD, Principal Investigator — University of California, San Diego; David R Murray, MD, Principal Investigator — University of Wisconsin, Madison; Amit Patel, MD, Principal Investigator — University of Utah Health Care, Utah
Locations (7):
- United States (7):
  - University of California, San Diego, San Diego, California
  - VA San Diego Healthcare System, San Diego, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Utah Health Care, Utah, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
The trial remains blinded

REFERENCES:
- [Derived] Hammond HK, Penny WF, Traverse JH, Henry TD, Watkins MW, Yancy CW, Sweis RN, Adler ED, Patel AN, Murray DR, Ross RS, Bhargava V, Maisel A, Barnard DD, Lai NC, Dalton ND, Lee ML, Narayan SM, Blanchard DG, Gao MH. Intracoronary Gene Transfer of Adenylyl Cyclase 6 in Patients With Heart Failure: A Randomized Clinical Trial. JAMA Cardiol. 2016 May 1;1(2):163-71. doi: 10.1001/jamacardio.2016.0008. PMID 27437887